CLINICAL TRIAL: NCT00611208
Title: A Phase II Study of A-dmDT390-bisFv(UCHT1) Fusion Protein in Patients With Cutaneous T Cell Lymphoma
Brief Title: A-dmDT390-bisFv(UCHT1) Immunotoxin Therapy for Patients With Cutaneous T-Cell Lymphoma (CTCL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Angimmune LLC (Industry)
Collaborators: James Graham Brown Cancer Center (Other); M.D. Anderson Cancer Center (Other); Scott and White Hospital & Clinic (Other); University of Texas Southwestern Medical Center (Other); Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDA IND 100712
Record Dates: First submitted 2008-01-25; First posted 2008-02-08 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: T-cell Lymphomas; T-cell Leukemia; Sezary Syndrome; Mycosis Fungoides; Cutaneous T-cell Lymphoma (CTCL)
MeSH Terms: conditions — Lymphoma, T-Cell; Leukemia, T-Cell; Sezary Syndrome; Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous | interventions — A-dmDT390-bisFv(UCHT1) protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A-dmDT390-bisFv(UCHT1) (Experimental): anti-T cell immunotoxin (antibody targeting CD3 on T-cells tagged with diptheria toxin)
  Interventions: Biological: A-dmDT390-bisFv(UCHT1)

INTERVENTIONS:
Biological: A-dmDT390-bisFv(UCHT1) — A-dmDT390-bisFv(UCHT1) will be administered as 60 μg/kg total given as 7.5 μg/kg/injection twice a day 4-6 hours apart for four consecutive days (days 1-4) into a free flowing IV over a period of approximately 15 minutes
  Other Names: Resimmune®

SUMMARY:
This is a Phase II clinical trial aimed at treating a subgroup of patients with cutaneous T-cell lymphoma. The drug consists of a toxin, called diphtheria toxin, which is attached to an antibody that can specifically target cancerous T-cells. Our primary objectives are, therefore, to determine the patient subgroup with respect to disease burden who best responds to this experimental drug in treating CD3 positive T cell malignancies. We will be determining how the patient and their disease respond to this research agent.

The Clinical Response Data analysis from October 2014 done at the completion of the Phase I portion of A-dmT390-bisFv(UCHT1) fusion protein clinical trial showed that there were 25 evaluable patients who received all 8 doses varying between 2.5 and 11.25 µg/kg per dose. There were responses at all the lower dose levels up to 7.5 µg/kg per dose. The overall response rate was 36% and the complete response rate was 16% (when followed for 6 months). We have identified a subgroup of CTCL patients that have a very high response rate. If we exclude patients whose mSWAT scores never exceeded 50 (50% of skin surface area times a multiplier) and who never had lymph node involvement or stage III disease we are left with 9 patients. This subgroup has an overall response rate of 89% and a complete response rate of 50% (when followed for 6 months). Of these 4 patients currently in complete remission, three are long-term responders. Two are over 6 years in duration and one over 5 years duration. These may represent cures. The long time periods in the transition from partial response to complete response without treatment, 6 months to two years, suggests that the study drug in addition to exerting a direct killing effect on tumor also functions as an immunomodulator.

DETAILED DESCRIPTION:
The purpose of this study is to further evaluate the clinical responses including response rate and duration and correlate with patient disease stage, tumor burden, anti-DT titer and degree of T cell depletion induced by A-dmDT390-bisFv(UCHT1) fusion protein for patients with surface CD3+ malignant diseases. The secondary objective is to further explore the toxicity profile of A-dmDT390-bisFv(UCHT1) fusion protein for a high-response subgroup of patients with CTCL whose disease stage has not progressed beyond stage IB/IIB with mSWAT < 50%. Patients will receive full supportive care including transfusions of irradiated washed blood and blood products, antibiotics, antiemetics, etc, when appropriate. However, other anti-neoplastic drugs or hematopoietic growth factors (e.g., erythropoietin, interleukin-11, G-CSF and GM-CSF) are not allowed. Treatment will consist of one 4 day cycle consisting of 2 daily infusions for a total of 8 treatments given on an outpatient basis. Patients will be monitored until day 14 for signs of late drug toxicity by a daily phone call from their health care provider. Subjects will be instructed on how to monitor their own blood pressure at home and encouraged to measure and chart their daily weights that they can report to their health care provider. Off-treatment follow-up will be based upon response. Patients who experience a partial or complete remission who later relapse can receive radiation treatment of new lesions and remain on study as this course is typical of responses to an immunomodulating drug. Patients will have a follow-up visit and testing on day 37. Patients with partial or complete remissions will have another follow-up visit on day 60, then every three months for 1 year, followed by annual visits to assess duration of the response. To accommodate patients, we are offering a travel reimbursement program. Due to the 4 days of consecutive infusions, we will reimburse the expense the patient would incur to travel to the participating institution for treatment.

Objectives:

1. Evaluate the overall clinical responses including response rate and duration in a larger group of CTCL high-response patients to see if is higher than current therapies (>49%).
2. Determine the complete response rate and duration of response of A-dmDT390-bisFv(UCHT1) fusion protein in a larger group of CTCL high-response patients to see if is higher than current therapies (>20%).
3. Further define toxicities of A-dmDT390-bisFv(UCHT1) regimen in patients with CTCL who have been selected to be free from preexisting cardiac disease and never treated with Campath.
4. Determine if correlations exist between disease stage, tumor burden, anti-DT titer and degree of T cell depletion and response rate and response duration.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have signed the current Institutional Review Board (IRB) approved informed consent prior to registration (see Informed Consent).
* All patients must have CTCL diagnosed by morphologic, histochemical or cell surface marker criteria with stage never exceeding IB / IIB disease and mSWAT < 50%. CTCL patients with stage IA disease are not eligible for enrollment. CTCL patients with stage IB disease are eligible provided that they have failed a systemic treatment (this includes radiation). CTCL patients with bone marrow involvement but without lymph node involvement are eligible. Patients with a diagnosis of angioimmunoblastic T cell lymphoma are eligible, even with lymph node involvement. Age ≥ 18 years. Patients must have a performance status of < 2 on Eastern Cooperative Oncology Group scale (see Appendix). Patients must have fully recovered from toxicity of prior chemotherapy or radiation therapy.
* Patients must have bilirubin < 1.5 mg/dL, transaminases < 2.5 X ULN, albumin > 3 gm/dL, creatinine < 2.0 mg/dL. Patients who have had albumin < 3 gm/dL boosted by an albumin infusion must be observed to maintain albumin at > 3gm dL for 30 days without an additional infusion.
* Patients must have a normal echocardiogram (EF > 50% normal) without any evidence of cardiac chamber hypertrophy, dilatation or hypokinesis. The Sponsor must be provided with copies of these tests BEFORE Sponsor will approve enrollment. In addition, the sponsor must receive a list of current medications taken by the patient before Sponsor will approve enrollment.
* Females and males must be willing to use an approved form of birth control while on this study and for 2 weeks after completion.

Exclusion Criteria:

* Failure to meet any of the criteria set forth in Section 3.1.
* Inability to give informed consent because of psychiatric problems, or complicated medical problems.
* Allergic to diphtheria toxin a component of the study drug A-dmDT390-bisFv(UCHT1).
* Serious concurrent medical problems, uncontrolled infections, or disseminated intravascular coagulopathy (DIC), hepatic cirrhosis, or chronic kidney disease.
* CNS leukemia.
* Preexisting cardiovascular disease. The only exception being well controlled essential hypertension with a sitting blood pressure (B.P.) of < 160 systolic and < 90 diastolic without any evidence of structural heart disease or one episode of myocardial infarction > 8 months ago. A past history of any of the following conditions is considered as exclusions to study participation:

  * Congestive heart failure,
  * Atrial fibrillation,
  * Pulmonary hypertension,
  * Anticoagulant drug therapy,
  * Thromboembolic events,
  * Cardiomyopathy or a myocardial infarction within the past 8 months.
  * The PI and the Clinical Coordinator will be asked to verify that their referred patients do not have these exclusionary histories listed in 3.2 and a copy of this verification must be sent to the Sponsor before the Sponsor will approve of enrollment. Referring physicians will not need to sign. (Template for verification letter Appendix C).
* Pregnant or nursing women will be excluded from study.
* History of cirrhosis of the liver based on the Child-Pugh score of Class B or C are not eligible to participate. (Appendix B.)
* Prior treatment with alemtuzumab (Campath) or similar agents or procedures that depress blood T cell counts to below 50% of the lower limit of normal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-01; Primary Completion 2015-02 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Remission status (complete, partial, stable disease, progressive disease) | Time Frame: 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Arthur E Frankel, MD, Principal Investigator — University of Texas Southwestern Medical Center; Madeleine Duvic, MD, Principal Investigator — M.D. Anderson Cancer Center; Cesar Rodriguez, MD, Principal Investigator — James Graham Brown Cancer Center
Locations (5):
- United States (5):
  - Yale University School Of Medicine Recruiting, New Haven, Connecticut
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Scott and White Hospital & Clinic, Temple, Texas

REFERENCES:
- [Result] Frankel AE, Zuckero SL, Mankin AA, Grable M, Mitchell K, Lee YJ, Neville DM, Woo JH. Anti-CD3 recombinant diphtheria immunotoxin therapy of cutaneous T cell lymphoma. Curr Drug Targets. 2009 Feb;10(2):104-9. doi: 10.2174/138945009787354539. PMID 19199905
- [Result] Frankel, Arthur E. Anti-CD3 immunotoxin to induce remissions in cutaneous T-cell lymphoma patients. Poster session presented at: 2012 American Society of Clinical Oncology (ASCO). Oral Abstract Session, Developmental Therapeutics - Clinical Pharmacology and Immunotherapy. 2012 June 1-5; Chicago, IL.
- [Result] Arthur E. Frankel, Jung H. Woo, Jeremy P. Mauldin, Francine M. Foss, Madeleine Duvic, David M. Neville Jr. An Update On The Clinical Activity Of Resimmune, a Targeted Therapy Directed To CD3 Receptor, In Patients With Cutaneous T Cell Lymphomas-CTCL. Poster session presented at: 2012 American Society of Hematology (ASH). 55th ASH Annual Meeting and Exposition. 2013 December 7-10; New Orleans, LA.
- [Result] Frankel AE, Woo JH, Ahn C, Foss FM, Duvic M, Neville PH, Neville DM. Resimmune, an anti-CD3epsilon recombinant immunotoxin, induces durable remissions in patients with cutaneous T-cell lymphoma. Haematologica. 2015 Jun;100(6):794-800. doi: 10.3324/haematol.2015.123711. Epub 2015 Mar 20. PMID 25795722
- See also: ASH 2013 Abstract — https://ash.confex.com/ash/2013/webprogram/Paper57379.html